CLINICAL TRIAL: NCT05059925
Title: Compare the Effects of Structured Gym Activities and Traditional Aerobic Activities in People With Cardiac Conditions
Brief Title: Structured Gym Activities and Aerobic Activities in People With Cardiac Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/01084 Anam Saif
Record Dates: First submitted 2021-09-18; First posted 2021-09-28 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Disease
Keywords: Gym Activities; Aerobic Exercises
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured gym activities (Experimental): Planned and structured activities such as Strength training for 4 weeks
  Interventions: Other: Structured gym activities
- Traditional aerobic activities (Active Comparator): Activities performed such as Treadmill , Cycle ergometer , Elliptical exercises for 4 weeks
  Interventions: Other: Traditional aerobic activities

INTERVENTIONS:
Other: Structured gym activities — Planned and structured activities such as Strength training
  * Dumbbell Exercises (1kg with 2 sets of 10 repetitions)
  * Sit-ups (2 sets of 10 repetitions)
  * Stair climbing, (2 sets of 10 stairs up and down)
  * Squat (2 sets of 10 repetitions) Flexibility training • Tai chi (Peng. Lu, chi, an Tsai, lieh, chou, Kao (Hold each posture for 20 seconds)) • Pilates (Breathing., Shoulder bridge, Leg lifts (Hold each pose for 20 seconds)) • Stretching techniques (Neck stretch, Shoulder stretch, Side stretch Hold each stretch for 20 seconds)).
  Arms: Structured gym activities
Other: Traditional aerobic activities — Activities performed such as
  * Treadmill Time: 10 minutes Intensity: 60 to 80% of target heart rate
  * Cycle ergometer Time: 10 minutes Intensity: 60 to 80% of target heart rate
  * Elliptical exercises Time: 10 minutes Intensity: 60 to 80% of target heart rate
  Arms: Traditional aerobic activities

SUMMARY:
To compare the effect of structured gym activities and traditional aerobic activities on cardiorespiratory endurance in people with cardiac conditions To compare the effect of structured gym activities and traditional aerobic activities on quality of life in people with cardiac conditions

ELIGIBILITY:
Inclusion Criteria:

* Individuals with cardiac conditions including post-first myocardial infarction, post valvular diseases, post-CABG patients.
* Individuals who can perform cardiorespiratory exercises with ease(who are able to complete 6 minute walk test).
* Individuals who have not performed regular physical activity in the past 6 months (PA-R)
* No regular exercise or gym activity since last 6 months

Exclusion Criteria:

* Individuals who are highly trained in gymnastic
* Already trained (any gym activity or regular exercise)
* Individuals with Diabetes, hypertension, and kidney diseases.
* Any neurological complication
* Any Musculoskeletal Disorder

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life SF-36 questionnaire | Changes from the baseline to 4th Week
  The Short Form 36 Health Survey Questionnaire (SF-36) questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). A final item, termed self-reported health transition, is answered by the client but is not included in the scoring process.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Oxygen Saturation (SpO2) | 4th Week
  Changes from baseline SPO2 was measured in percentage. Oxygen immersion is the division of oxygen-soaked hemoglobin with respect to add up to hemoglobin in the blood. Pulse oximeter measure it.
Pulse Rate | 4th Week
  Changes from baseline, Pulse rate was measured per minute through pulse oximeter
Modified Borg Scale of Perceived Exertion | 4th week
  Changes from the Baseline, It is a subjective numeric scale ranging from 0 to 10, where 0 indicates "no dyspnea" and 10 indicates "unbearable dyspnea." A number is chosen by the patient in order to decide the best score that matches his level of dyspnea during physical activity.
Systolic and diastolic blood pressure | 4th week
  Changes from the Baseline, Blood pressure is measured through sphygmomanometer
VO2 max | 4th week
  Changes from the Baseline, Maximal oxygen consumption (VO2 max), refers to the maximum amount of oxygen that an individual can utilize during intense or maximal exercise.
METS | 4th Week
  Changes from the Baseline, Metabolic equivalents (METS) Associated with Common Types of Endurance Exercise.
  METs may be calculated during Standard Bruce Protocol by dividing oxygen uptake per minute with the product of 3.5 × bodyweight (kilograms)
Quick Physical Activity Rating (QPAR) scale | 4th Week
  10 items covering passive activities, walking, hobby and recreational activities, exercise, and housework with exemplars provided. Hobby activities, exercise and housework were further divided into light, moderate, and strenuous activities. Respondents were asked to consider these physical activities over the prior 4-week period. Each activity was weighted in intensity ranging from 1 (light) to 3 (heavy) intensity. Frequency of activity per week was collected as never (0 days), seldom (1-2 days), sometimes (3-4 days), and often (5-7 days). Duration of activity was collected as less than one hour per day, 1-2 hours per day, and more than two hours per day. Multiplication of the intensity (1-3), frequency (0-3) and duration (1-3) scores permitted calculation of a dose of physical activity ranging from 0-153. The QPAR took 3-5 minutes to complete. Changes from the baseline to 4th week

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Fitlytics gym Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No